CLINICAL TRIAL: NCT06464263
Title: Comparative Study Between Dexmedetomidine Versus Midazolam-Fentanyl for Analgesia and Sedation After Adult Valvular Cardiac Surgeries; a Prospective Randomized Blinded Clinical Trial
Brief Title: Dexmedetomidine Versus Midazolam-Fentanyl for Analgesia and Sedation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anesth-._098/2023
Record Dates: First submitted 2024-06-09; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Valvular Cardiac Surgeries
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): This Group about 30 patients will receive a loading dose of 1 μg/kg dexmedetomidine (Precedex 4 mcg/ml, Pfizer. Inc, New York, USA) diluted in 100 ml 0.9% saline infused over 10 min immediately postoperative, followed by continuous infusion of 0.2-0.7 μg/kg/h.
  Interventions: Drug: Dexmedetomidine
- Fentanyl Group (Experimental): This Group about 30 patients will receive an initial bolus dose of fentanyl (fentanyl 50 mcg/ml, hameln; Netherlands) of 1-2 μg/kg, followed by an infusion at an initial rate of 1 to 2 μg/kg/h.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — to investigate the postoperative analgesic-sedative effect of dexmedetomidine versus fentanyl-midazolam to achieve fast-track extubation after adult valvular cardiac surgeries.
  Other Names: fentanyl 50 mcg/ml

SUMMARY:
Postoperative sedation is an essential component in recovery of the patient undergoing cardiac surgery. It facilitates the patient's unawareness of the environment as well as reduce the discomfort and anxiety caused by surgery, intubation, mechanical ventilation, suction, and physiotherapy.

Despite the advances in anesthesia and surgical techniques, the duration of mechanical ventilation (MV) may be prolonged after cardiac surgery, due to the classic high-dose narcotic-based cardiac anesthesia.

DETAILED DESCRIPTION:
In recent years, fast-track extubation (FTE) protocols have been developed to reduce the long period of intubation and complications that may occur due to the long duration of MV. Potential advantages of FTE protocols following surgery for congenital cardiac disease are reduced ventilator-associated pulmonary complications and the negative effects of positive pressure ventilation, reduced nosocomial infections, postoperative atelectasis, reduced requirements of sedatives and analgesic drugs, early enteral feeding, rapid patient mobilization, and shorter intensive care unit (ICU) stay.

The ideal analgesic-sedative agents would keep the patient comfortable without anxiety. It would effectively provide adequate sedation, but also allow neurologic evaluation of the patient, ideally without stopping administration of the drug. It would have minimal hemodynamic and respiratory depressant effects. It also would have a rapid onset and offset of action without drug accumulation or active metabolites, making it easily titratable and allowing rapid recovery with a prompt return to normal activity after discontinuation.

Opioids and benzodiazepines are the most frequently used analgesic-sedative agents after cardiac surgery. Although opioid can provide excellent analgesia, the doses for effective pain relief may lead to undesirable side effects, such as respiratory depression requiring prolonged MV, hemodynamic instability, tolerance, and significant withdrawal symptoms that also delay patient recovery.

Dexmedetomidine is a highly selective α2-adrenoreceptor agonist. Presynaptic activation of α2-adrenoreceptors at sympathetic nerve endings inhibits catecholamine release. The major effect of dexmedetomidine is maintaining sedation-analgesia without a respiratory depressant effect. It has relatively few cardiovascular side effects and produces sleep-like sedation without narcosis or respiratory depression.

Indeed, current guidelines recommend lighter levels of sedation to manage ventilated patients preferably using nonbenzodiazepine sedatives. Nevertheless, there is currently no consistent recommendation regarding which nonbenzodiazepine sedative agents should be used.

ELIGIBILITY:
Inclusion Criteria:

- This study will include patients undergoing elective adult valvular cardiac surgeries

Exclusion Criteria:

* Patient refusal.
* Emergent valve cardiac surgeries.
* Patients with known hypersensitivity to study drugs.
* History of uncontrolled diabetes or hypertension.
* Impaired kidney or liver functions.
* Perioperative hemodynamic instability.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Pain Relieve | 2 hours post operative
  Assessment of the pain post-operatively in patients with pain score by VAS as : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ibrahim Mohammed Hashish, Professor, Study Chair — Al-Azhar University, Faculty of medicine; Mohamed husseiny Mahmoud, Lecturer, Principal Investigator — Cardio-Thoracic Surgery Department, Al-Azhar University
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided